CLINICAL TRIAL: NCT01033110
Title: Fit Over 45 - a Health Promotion Project for Inactive Female Hospital Staff Age 45+ From the University Hospital of Zürich
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-bischoff
Record Dates: First submitted 2009-11-25; First posted 2009-12-16 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: inactive; >45 years; female
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise; Nutrition Assessment

INTERVENTIONS:
Behavioral: Exercise and Nutrition Education — Guided nordic walking training and 12 presentations about diet and health.

SUMMARY:
Background:

Despite the well-known benefits of exercise, 64% of the Swiss population do not fulfill the public health recommendation of physical activity. A survey of female staff members over 45 years of age from the University Hospital Zurich at the end of 2003 showed that physical inactivity is also prevalent in this population.

Aim:

To assess whether inactive women working at a large hospital centre prefer Nordic Walking (NW) or a Jogging (J) as a health promotion strategy. (2) To test whether the method chosen by the majority improves physical performance, physical activity, body weight and composition, and bone mineral density.

Methods: The investigators will send out a questionnaire to all female staff members at a large hospital centre age 45 and older, ask whether they are inactive, and whether they prefer Nordic Walking or Jogging as a health promotion strategy. Depending on the preference of the majority of the women, the investigators will then ask inactive female staff members age 45+ to participate in a 12-months randomized controlled trial comparing training plus nutrition education to nutrition education alone. The training will have a 3-month building-up phase followed up by an in part unsupervised training of 9 months. All participants will receive a lecture on healthy nutrition once a months for 12 months. The investigators will assess diet with a food frequency questionnaire at baseline and after 12 and 24 months.

The primary endpoint is: physical performance, measured with the 12-minute Coopertest.

The secondary endpoints are: level of physical activity, body mass index, body composition and bone mineral density at the spine and the hip.

Importance: This project will address the questions which physical activities are preferred by inactive women and whether the preferred training improves physical performance, physical activity, body mass index, body composition and bone mineral density. In addition, our study will explore whether those women who changed their diet in addition to being randomized to the training group have an enhanced benefit.

ELIGIBILITY:
Inclusion criteria:

* USZ-staff, at least 45 years old, insufficiently active according to the Swiss recommendation of health enhancing physical activity (neither 30 minutes of moderate physical activity at least five days in the week nor 20 minutes of vigorous physical activity at least two times per week) and written informed consent.

Exclusion criteria:

* Acute osteoporotic fracture (<3 month), disability of the musculoskeletal system or cardiovascular diseases which do not allow an endurance training.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
physical performance | baseline, 3, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff Ferrari, MD, MPH, Principal Investigator — University Hospital Zurich, Centre on Aging and Mobility
Locations (1):
- University Hospital Zurich, Centre on Aging and Mobility, Zurich, Canton of Zurich, Switzerland